CLINICAL TRIAL: NCT06683781
Title: Ventilatory Settings and Monitoring Variables Associated With Weaning Failure in Critically Ill Patients: A Retrospective Study
Brief Title: Ventilatory Settings and Monitoring Variables Associated With Weaning Failure in Critically Ill Patients
Acronym: WEAN-FAIL
Status: Recruiting | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, EMILIO MARTIN STEINBERG, Principal Investigator, Hospital Italiano de Buenos Aires
Other Study IDs: 7221
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Mechanical Ventilation; Weaning Failure; Weaning Failure of Mechanical Ventilation; Intensive Care Unit ICU
Keywords: weaning failure; mechanical ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically ventilated patients

SUMMARY:
Mechanical ventilation (MV) is essential in managing acute respiratory failure. Its duration is a crucial aspect since both, unnecessary prolongation and premature withdrawal have deleterious effects on patient outcomes in the ICU. The process of weaning refers to the set of procedures and evaluations carried out to discontinue MV. Regardless of the definition used, within the population undergoing weaning, there is a group of patients who successfully pass the daily screening but fail the spontaneous breathing trial (SBT) or the separate attempt (SA). In Argentina, this figure is 39.5%, and 31.4% in patients with COVID-19. On the other hand, another group of patients successfully passes the SA, is extubated, but fails in post-extubation. This failure rate varies in the literature, ranging from approximately 10 to 20%. In our country, this figure is 16% in the general population and rises to 29.7% in COVID-19 patients. Additionally, this population is divided into those who cannot tolerate ventilation without an artificial airway due to upper airway patency issues (such as laryngeal edema), i.e., "airway failure," and those who experience acute respiratory failure. In 2023, the WEAN SAFE study reported novel findings regarding variables associated with weaning failure. In multivariable analysis, it was found that the MV settings and monitoring variables at the time of the first SBT - respiratory rate, positive end-expiratory pressure (PEEP), dynamic airway pressure difference (peak pressure (Ppeak) minus PEEP) on the day of the SA - were associated with weaning failure. In this context, the investigators will conduct a retrospective cohort study, whose primary objective will be to assess which MV settings and monitoring variables are associated with weaning failure.

**Primary Objective** To determine if there are any MV settings or monitoring variables that are associated with extubation failure.

**Secondary Objective** To determine if there are any MV settings or monitoring variables that are associated with failure in the first SBT.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* MV for at least 48 hours, regardless of the cause of onset
* Undergone at least one extubation, regardless of the outcome
* At least one spontaneous breathing trial (SBT) during their ICU stay, regardless of the outcome

Exclusion Criteria:

* MV records containing incorrect or inconsistent data
* did not have adequate or continuous monitoring during the weaning process

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients who required MV and underwent a weaning process in the ICU admitted up to July 1, 2024, whose MV settings and monitoring data are complete in their medical records.
Sampling Method: Probability Sample
Enrollment: 1077 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with extubation failure | 7 days
  Need for reintubation within the first 7 days after the removal of the endotracheal tube, regardless of the cause that precipitates it.
Cause of reintubation | 7 days
  Reason that precipitates the need for reinsertion of the endotracheal tube.

SECONDARY OUTCOMES:
Spontaneous breathing trial failure | Immediately after spontaneous breathing trial
  Rate of restoring invasive MV due to objective or subjective signs.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No